CLINICAL TRIAL: NCT00342030
Title: Dietary and Genetic Factors in Asthma & Chronic Bronchitis in a Cohort of Chinese Singaporeans
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903044; 03-E-N044
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-12

CONDITIONS: Chronic Bronchitis; Asthma
Keywords: Respiratory; Polymorphism; Fruit; COPD; Prospective; Diet
MeSH Terms: conditions — Bronchitis, Chronic; Asthma; Pulmonary Disease, Chronic Obstructive

SUMMARY:
There is suggestive evidence for a role of dietary in the etiology of asthma and chronic bronchitis. However, there are few prospective data. We propose to expand our collaboration with the Singapore Chinese Health Study to examine dietary, environmental, and genetic factors, along with their interactions, in relation to the risk of developing asthma and chronic bronchitis. The Singapore Chinese Health Study is a cohort of 63,257 men and women of Chinese ethnicity in Singapore who were aged 45-74 years at enrollment from 1993 to 1998. Telephone follow-up of the cohort to update and outcome information began in 1999 and is ongoing. We expect to identify 538 cases of incident asthma and 672 cases of incident chronic bronchitis when the current follow-up questionnaire cycle is complete in 2004. In this proposal, we would validate self-reports of incident asthma, obtain follow-up data from the entire cohort to perform analyses of dietary and smoking in relation to these outcomes, and analyze genetic material on cases of incident asthma and chronic bronchitis and controls from the cohort. In this proposal we will examine the following hypotheses:

1. Higher intake of fruits and/or antioxidant micronutrients decreases the risk of developing asthma and chronic bronchitis.

   a. Effects if fruit and/or antioxidant micronutrients may differ by smoking history.
2. Common polymorphisms in genes involved in the response to oxidative stress influence the risk of asthma and chronic Bronchitis. We initially propose to examine polymorphisms in three genes--glutathione S-tranferase M1, glutahione S-transferase P1, and matrix metalloproteinase-1. However, we plan to examine additional relevant polymorphisms in the future, especially taking advantage of high throughput screens of candidate genes for asthma and chronic bronchitis. It is possible that by 2004 when the sample set will be available that more compelling candidates and high throughput screens may be available to us at a low cost. Thus we will re-evaluate our choice when the samples are available.
3. Polymorphisms in these and other genes interact with fruit/antioxidant intake and/or smoking to influence the risk of asthma and chronic bronchitis.

DETAILED DESCRIPTION:
There is suggestive evidence for a role of diet in the etiology of asthma and chronic bronchitis. However, there are few prospective data. We propose to expand our collaboration with the Singapore Chinese Health Study to examine dietary, environmental, and genetic factors, along with their interactions, in relation to the risk of developing asthma and chronic bronchitis. The Singapore Chinese Health Study (NIH grant CA080205) is a cohort of 63,257 men and women of Chinese ethnicity in Singapore who were aged 45-74 years at enrollment from 1993 to 1998. Telephone follow-up of the cohort to update and outcome information began in 1999 and is ongoing. We expect to identify 538 cases of incident asthma and 672 cases of incident chronic bronchitis when the current follow-up questionnaire cycle is complete in 2004. In this proposal, we would validate self-reports of incident asthma, obtain follow-up data from the entire cohort to perform analyses of diet and smoking in relation to these outcomes, and analyze genetic material on cases of incident asthma and chronic bronchitis and controls from the cohort. In this proposal we will examine the following hypotheses:

1. Higher intake of fruits and/or antioxidant micronutrients decreases the risk of developing asthma and chronic bronchitis.

   a. Effects of fruit and/or antioxidant micronutrients may differ by smoking history
2. Common polymorphisms in genes involved in the response to oxidative stress influence the risk of asthma and chronic bronchitis. We initially propose to examine polymorphisms in three genes -- glutathione S-tranferase M1, glutathione S-transferase P1, and matrix metalloproteinase-1. However, we plan to examine additional relevant polymorphisms in the future, especially taking advantage of high throughput screens of candidate genes for asthma and chronic bronchitis. It is possible that by 2004 when the sample set will be available that more compelling candidates and high throughput screens may be available to us at a low cost. Thus we will re-evaluate our choice when the samples are available.
3. Polymorphisms in these and other genes interact with fruit/antioxidant intake and/or smoking to influence the risk of asthma and chronic bronchitis.

ELIGIBILITY:
* INCLUSION CRITERIA:

No new subjects are being enrolled for this proposal.

Subjects are the 63,257 participants in the Singapore Chinese Health Study. That study includes men and women aged 45-74 at enrollment of Chinese ethnicity living in Singapore.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63257 (Estimated)
Dates: Start 2002-11-01; Study Completion 2012-04-12

CONTACTS AND LOCATIONS:
Overall Officials: Frederick W Miller, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- National University of Singapore, Kent Ridge, Singapore

REFERENCES:
- [Background] Buist AS, Vollmer WM. Reflections on the rise in asthma morbidity and mortality. JAMA. 1990 Oct 3;264(13):1719-20. No abstract available. PMID 2398613
- [Background] Ng TP, Hui KP, Tan WC. Prevalence of asthma and risk factors among Chinese, Malay, and Indian adults in Singapore. Thorax. 1994 Apr;49(4):347-51. doi: 10.1136/thx.49.4.347. PMID 8202905
- [Background] Karjalainen A, Kurppa K, Martikainen R, Klaukka T, Karjalainen J. Work is related to a substantial portion of adult-onset asthma incidence in the Finnish population. Am J Respir Crit Care Med. 2001 Aug 15;164(4):565-8. doi: 10.1164/ajrccm.164.4.2012146. PMID 11520716